CLINICAL TRIAL: NCT05056961
Title: Effects of Large Tidal Volumes Despite Minimal Inspiratory Support in Spontaneously Ventilated Intubated Resuscitation Patients. Pathophysiological Exploratory Study.
Acronym: InLarge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: InLarge (RBHP 2018 Godet 2)
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Invasive Mechanical Ventilation; Ventilator-Induced Lung Injury; Patient-Self Inflicted Lung Injury; Encephalopathy; Intensive Care Unit; Tidal Volume
Keywords: ICU; Mechanical Ventilation; Ventilator-Induced Lung Injury; Patient-Self Inflicted lung Injury; Tidal volume
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Brain Diseases

STUDY DESIGN:
Intervention Model Description: Two parallel groups
  1. the first without respiratory distress symptoms
  2. the second with respiratory distress symptoms (for example, supra-clavicular and thoracic-abdominal asynchronies...)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large tidal volumes without respiratory distress symptoms (Other): Large tidal volumes (> 10 mL.kg-1 of predicted body weight) despite low pressure support, without respiratory distress symptoms
  Interventions: Other: Multiparametric mesurements
- Large tidal volumes with respiratory distress symptoms (Other): Large tidal volumes (> 10 mL.kg-1 of predicted body weight) despite low pressure support, with respiratory distress symptoms (for example, supra-clavicular and thoracic-abdominal asynchronies...)
  Interventions: Other: Multiparametric mesurements

INTERVENTIONS:
Other: Multiparametric mesurements — Multiparametric assessments will necessitate the use of a plastic belt to record electro-impedancemetry tomography data; and a nano-gatsric tube fitted with esophageal and gastric low pressure balloons
  Other Names: Oesophageal pressure; Gastric pressure; P0,1; Tomography electro-impedancemetry

SUMMARY:
Some ICU ventilated patients might present with large tidal volume despite very low or inexistant presser support. Patient-Self Inflicted Lung Injury (P-SILI) might appear related with large alveolar stretch an distension. Two clinical presentations are observed: patients with or without respiratory distress signs such as supra-clavicular depression and thoracic-abdominal asynchronies.

The aim of this study is to compare the pulmonary physio(-patho)logical parameters of these two types of patients (eupneic or with respiratory distress signs), and presenting important TV in spite of a minimal adjustment of the ventilatory support, except for Acute Respiratory Distress Syndrome (ARDS).

DETAILED DESCRIPTION:
The use of invasive mechanical ventilation is one of the most frequent therapies in the intensive care unit. There are several types of indication, depending on the failure: mainly neurological, hemodynamic or respiratory. In recent years, the concept of Ventilator Induced Lung Injury (VILI) has led to changes in ventilator settings in both intensive care units and operative rooms. Thus, tidal volume (TV) reduction to 6-8 mL.kg-1 of predicted body weight, the use of an individualized positive end-expiratory pressure (PEEP) and the possible use of therapies to optimize pulmonary aeration (alveolar recruitment maneuvers, prone positioning sessions...) have become mandatory. More recently, some authors have described the existence of Patient-Self Inflicted Lung Injury (P-SILI). In certain situations (delirium, encephalopathies, pulmonary receptor stimulation, metabolic acidosis...), some patients may present, in spite of an "optimized" ventilator setting, very important VT, which may exceed 10 mL.kg-1 of theoretical ideal weight. Two circumstances of observation of these large VT needs despite low pressure supports can be observed. The first corresponds to a patient with signs of respiratory distress (signs of respiratory distress: supra-clavicular, thoraco-abdominal asynchronies...) who presents with significant inspiratory efforts. The second is a patient with no sign of respiratory distress (eupnea). In both cases, the "trigger" comes from a (hyper)-stimulation (drive) of respiratory brainstem centers.

It is currently uncertain whether these two types of patients are comparable in terms of P-SILI. It is possible that in the second case, lesions are non-existent (or minimal) due to low trans-pulmonary pressure (stress) and low levels of pulmonary alveolar distension (strain). Indeed, the most likely determinant of alveolar injury is trans-pulmonary pressure, defined as the difference between upper airway pressure and pleural pressure (Ptp = Paw - Ppl). Thus, in case of a negative pathophysiological parameter, it would be preferable to sedate the patient more deeply and to temporarily consider controlled mechanical ventilation to limit the alveolar stretch and lesions. However, we know that excessive sedation of resuscitation patients increases their morbidity and mortality, by exposing them to increased duration of mechanical ventilation, and thus to the risk of pneumonia acquired under mechanical ventilation. In this context, daily sedation release tests are recommended. Physicians must therefore find the right balance between an optimal level of sedation compatible with the least deleterious ventilatory support possible.

The aim of this study is to compare the pulmonary physio(-patho)logical parameters of these two types of patients (eupneic or with respiratory distress signs), and presenting important TV in spite of a minimal adjustment of the ventilatory support, except for Acute Respiratory Distress Syndrome (ARDS).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients admitted to the adult intensive care unit at Estaing Hospital, Clermont-Ferrand
* Patients under invasive mechanical ventilation (intubation or tracheostomy)
* Patients with a tidal volume greater than 10 mL.kg-1 of predicted body weight despite a minimal pressure support (< 5 cmH2O)
* Patients with sedation compatible with spontaneous ventilation with inspiratory support and positive end-expiratory pressure
* Patient calm (RASS between -2 and 0)
* Consent to participate in the study from the patient or authorization to carry out the research collected from the designated trusted person (failing that, a family member or a close relative who has a close and stable relationship with the patient) in accordance with the procedures described in Title II of the First Book of the Public Health Code. If no relative is present, the patient may be included on the advice of the investigator (article L. 1111-6). A consent form for the continuation of the study and the use of the data will then be signed by the patient if and when he/she is conscious and lucid again, or if the patient is unable to express his/her consent, an authorization to continue the research will be obtained from the designated trusted person
* Patient benefiting from a Social Security system

Exclusion Criteria:

* Refusal to participate in the proposed study
* Protected adults
* Contraindication to the placement of a nasogastric tube:

  * Severe uncorrected blood flow disorder
  * Known naso-sinusal lesion
  * Recently ligated esophageal varices (< 48h)
* Contraindication to the use of the tomographic electroimpedancemetry technique

  * Thoracic lesions
  * Thoracic dressings
  * Pace-maker/implantable defibrillator
* Known injury to central respiratory centers, including neurocompromised patients
* Patients with Acute Respiratory Distress Syndrome (according to Berlin criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-21 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-06-25 (Estimated)

PRIMARY OUTCOMES:
Transpulmonary driving pressure | During 1 hour starting from inclusion
  Comparison of transpulmonary motor pressure levels during spontaneous invasive mechanical ventilation of patients with large tidal volumes (>10 mL.kg-1 theoretical ideal weight) despite minimal pressure support (inspiratory support <5 cmH20). Transpulmonary motor pressure is defined as follows:
  ΔPtp = (Pplateau - Inspiratory Poeso) - (PEEP - Expiratory Poeso)

SECONDARY OUTCOMES:
Transpulmonary pressure (alveolar stress) | At inclusion and after 1 hour
  Maximum transpulmonary pressure (alveolar stress) defined as follows:
  Ptp = Pplateau - Inspiratory Poeso
Pressure of respiratory occlusion (P0,1) | At inclusion and after 1 hour
  Pressure of respiratory occlusion (P01) representative of respiratory drive, automatically delivered by the ventilator
Driving pressure | At inclusion and after 1 hour
  Driving pressure
Work of breathing | At inclusion and after 1 hour
  Work of breathing as defined as follows:
  WOB = ΔP x ΔV during inspiration
Alveolar strain | At inclusion and after 1 hour
  Alveolar strain defined as follows:
  Strain = TV / FRC
Energy transmitted to the patient's lungs by the ventilator | At inclusion and after 1 hour
  Energy transmitted to the patient's lungs by the ventilator as defined by Gattinoni et al. (Intensive Care Medicine 2016)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Clermont-Ferrand, France